CLINICAL TRIAL: NCT01939756
Title: Intravesical Natural Baobab Oil in the Management of BCG-induced Lower Urinary Tract Symptoms: a Phase I-II Study
Brief Title: Intravesical Natural Baobab Oil in the Management of BCG-induced Lower Urinary Tract Symptoms
Acronym: Baobab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Savino M. Di Stasi (Other)
Collaborators: University of Bari (Other)
Responsible Party: Sponsor-Investigator, Savino M. Di Stasi, Associate Professor of Urology, MD, PhD, University of Rome Tor Vergata
Organization: University of Rome Tor Vergata (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTV-101-2012
Record Dates: First submitted 2013-09-02; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Superficial Bladder Cancer; Lower Urinary Tract Symptoms
Keywords: High risk non-muscle invasive urothelial bladder cancer; Intravesical BCG; Local toxicity; Natural baobab oil
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravesical baobab oil (Experimental): Intravesical instillation of 50 ml sterile Baobab natural oil. After draining of the bladder, the suspension is infused intravesically through a Foley catheter. The solution is retained in the bladder for 60 min, followed by emptying of the bladder and removal of the catheter.
  Interventions: Device: Intravesical baobab oil

INTERVENTIONS:
Device: Intravesical baobab oil — Intravesical baobab oil
  Other Names: Baotrophic, Physion Srl, Mirandola, Italy

SUMMARY:
Baobab oil is often used in traditional medicine as antipyretic, antioxidant, anti-inflammatory, analgesic and antimicrobial. It also regenerates the epithelial tissue in a short time improving tone and elasticity. We want to evaluate the effects of intravesical Baobab oil in patients with BCG-induced lower urinary tract symptoms.

DETAILED DESCRIPTION:
After complete transurethral resection of primary high risk non-muscle invasive bladder tumors (stage pTa, pT1, carcinoma in situ and high grade urothelial carcinoma), patients on induction course of intravesical BCG with lower urinary tract symptoms unresponsive to standard therapies are enrolled. The patients supply written informed consent to a document describing the investigational nature of the protocol.

Induction treatment consists of an initial 6 intravesical BCG treatments at weekly interval commencing approximately 3 weeks after transurethral resection procedures. The BCG instillation consisted of 81 mg wet weight (10•2±9•0 x 108 colony-forming units) BCG Connaught substrain. Lyophilised (ie, freeze-dried) BCG is suspended in 50 mL bacteriostatic-free solution of 0•9% sodium chloride. After draining of the bladder, the suspension is infused intravesically through a Foley catheter. The solution is retained in the bladder for 120 min, followed by emptying of the bladder and removal of the catheter.

During BCG treatment patients with persistent lower urinary tract symptoms unresponsive to standard therapies (anticholinergics, alpha-blockers, antibiotics, analgesics and anti-inflammatory drugs) are treated with an intravesical instillation of 50 ml sterile Baobab natural oil (Baotrophic, Physion Srl, Mirandola, Italy). After draining of the bladder, the suspension is infused intravesically through a Foley catheter. The solution is retained in the bladder for 60 min, followed by emptying of the bladder and removal of the catheter.

Lower urinary tract symptoms are self-recorded by the patients before and after each baobab oil instillation and classified by the investigator according to a classification grid considering account duration and intensity. The classification of symptoms is class 0= none, class I = mild, class II = moderate, and class III = severe, according to severity. Local adverse events are cystitis, nocturia, pollakiuria, micturition urgency, micturition burning, stress urinary incontinence, dysuria, hematuria, pelvic pain, and perineal pain. The outcome measures are analyzed before and every day for one week after treatment. All patients are assessed for safety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Complete transurethral resection of primary histologically proven high risk urothelial non-muscle invasive bladder tumors: high grade (G3,) stage pTa, pT1, and carcinoma in situ (pTis
* Intravesical BCG treatment
* Adequate bone marrow reserve (ie, white-blood-cell count ≥4000 x106 cells/L and platelet count

  ≥120 x 109/L
* Normal renal function (function (ie, serum creatinine ≤123•76 µmol/L)
* normal liver function ((ie, serum glutamic-oxaloacetic transaminase ≤42 U/L, serum glutamic-pyruvic transaminase ≤48 U/L, and total bilirubin ≤22•23 µmol/L)
* Karnofsky performance score of 50 to 100

Exclusion Criteria:

* Previous intravesical treatment with chemotherapeutic and immunotherapeutic drugs
* Previous or concomitant urothelial carcinoma of the upper urinary tract and urethra, or both
* Previous muscle-invasive (ie, stage T2 or higher) urothelia carcinoma of the bladder
* Known allergy to baobab oil
* Bladder capacity less than 200 mL
* Untreated urinary-tract infection
* Severe systemic infection (ie, sepsis)
* Urethral strictures that would prevent endoscopic procedures and catheterisation
* Disease of upper urinary tract (eg, vesicoureteral reflux or urinary-tract stones) that would make multiple transurethral procedures at risk
* Previous radiotherapy to the pelvis;
* Other concurrent chemotherapy;
* Treatment with radiotherapy-response or biological-response modifiers;
* Other malignant diseases within 5 years of trial registration (except for basal-cell carcinoma);
* Pregnancy or nursing;
* Psychological, familial, sociological, or geographical factors that would preclude study participation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Quantitative symptom score questionnaire | 36 months
  A quantitative symptom score questionnaire is completed by the patients before treatment to establish baseline symptoms and daily during the following 7 days after treatment. The questionnaire is designed to evaluate 10 lower urinary tract symptoms (cystitis, nocturia, pollakiuria, micturition urgency, micturition burning, stress urinary incontinence, dysuria, hematuria, pelvic pain, and perineal pain. Most symptoms are scored on a 0 to 3-point scale, corresponding to none/mild/moderate/severe.

SECONDARY OUTCOMES:
Baobab oil toxicity | 36 months
  All patients are assessed for safety or allergy to intravesical baobab oil

CONTACTS AND LOCATIONS:
Overall Officials: Savino M Di Stasi, MD, PhD, Study Chair — Tor Vergata University, Rome, Italy
Locations (2):
- Italy (2):
  - Savino M. Di Stasi, Rome
  - Tor Vergata University, Rome